CLINICAL TRIAL: NCT00719056
Title: Efficacy of Teicoplanin for the Prevention of Surgical Site Infections After Total Hip or Knee Arthroplasty: A Prospective, Open-Label Randomized Study
Brief Title: Teicoplanin Prophylaxis for Total Hip or Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: KAT Hospital of Athens (Unknown)
Responsible Party: University of Athens, Medical School, Greece
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEICO01
Record Dates: First submitted 2008-07-14; First posted 2008-07-21 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Total Hip and Knee Arthroplasties
Keywords: teicoplanin; prophylaxis; arthroplasty; surgical site infections
MeSH Terms: conditions — Surgical Wound Infection | interventions — Teicoplanin; Glycopeptides; Ciprofloxacin; Cephalosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Surgical chemoprophylaxis of one dose of teicoplanin upon introduction of anesthesia for total hip or knee arthroplasty.
  Interventions: Drug: Teicoplanin
- 2 (Active Comparator): Surgical chemoprophylaxis with multiple dose of other antimicrobials for up to six consecutive days for total hip or knee arthroplasty.
  Interventions: Drug: β-lactams or ciprofloxacin

INTERVENTIONS:
Drug: Teicoplanin — The selected dose was 10mg/kg and it was given intravenously by a catheter inserted under aseptic conditions in a forearm vein within 15 minutes; it was diluted in one 5% glucose solution of a 50 ml final volume
  Other Names: Glycopeptide
  Arms: 1
Drug: β-lactams or ciprofloxacin — Multiple doses for up to six consecutive days
  Other Names: Cephalosporins or ciprofloxacin or penicillincs
  Arms: 2

SUMMARY:
This is a prospective, open-label, randomized clinical trial where patients were administered prophylaxis for total hip or knee arthroplasty either with teicoplanin or with other antibiotics. The study is aiming to evaluate any differences between these two different strategies of antimicrobial prophylaxis in the occurrence of surgical site infections

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized clinical trial where patients were administered prophylaxis for total hip or knee arthroplasty either with a single dose of teicoplanin or with multiple doses of other antibiotics according to the habits of the attending physicians aiming to evaluate any differences between these two different strategies of antimicrobial prophylaxis in the occurrence of surgical site infections

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for total hip arthroplasty
* Patients admitted for total knee arthroplasty

Exclusion Criteria:

* Revision arthroplasty
* History of any infection within the preceding two months
* History of an operation in the same hip or knee for other causes
* Known history of allergy to the studied drug
* Pregnancy or lactation
* Any antibiotic therapy in the week before operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2004-08; Primary Completion 2005-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of single dose teicoplanin compared with comparator agents in the prevention of surgical site infections after total hip or knee arthroplasty. | Two years

SECONDARY OUTCOMES:
To compare the efficacy of single dose teicoplanin compared with comparator agents in the separate prevention of superficial or deep surgical site infections after total hip or knee arthroplasty. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Helen Giamarellou, MD, PhD, Study Chair — 4th Department of Internal Medicine, University of Athens, Medical School, Greece; Amyntas Varvaroussis, MD, Principal Investigator — 3rd Department of Orthopedics, KAT Hospital, Maroussi, Greece; Panagiotis Papadelis, MD, Principal Investigator — 2nd Department of Orthopedics, KAT Hospital, Maroussi, Greece; Vassilios Nikolaidis, MD, Principal Investigator — 4th Department of Orthopedics, KAT Hospital, Maroussi, Greece; Antonios Papadopoulos, MD, PhD, Study Director — 4th Department of Internal Medicine, University of Athens, Medical School, Greece
Locations (3):
- Greece (3):
  - 2nd Department of Orthopedics, KAT Hospital, Marousi, Athens
  - 3rd Department of Orthopedics, KAT Hospital, Marousi, Athens
  - 4th Department of Orthopedics, KAT Hospital, Marousi, Athens

REFERENCES:
- [Background] Soriano A, Popescu D, Garcia S, Bori G, Martinez JA, Balasso V, Marco F, Almela M, Mensa J. Usefulness of teicoplanin for preventing methicillin-resistant Staphylococcus aureus infections in orthopedic surgery. Eur J Clin Microbiol Infect Dis. 2006 Jan;25(1):35-8. doi: 10.1007/s10096-005-0073-z. PMID 16424973
- [Background] Wilson AP, Gruneberg RN, Neu H. Dosage recommendations for teicoplanin. J Antimicrob Chemother. 1993 Dec;32(6):792-6. doi: 10.1093/jac/32.6.792. No abstract available. PMID 8144419
- [Background] Nehrer S, Thalhammer F, Schwameis E, Breyer S, Kotz R. Teicoplanin in the prevention of infection in total hip replacement. Arch Orthop Trauma Surg. 1998;118(1-2):32-6. doi: 10.1007/s004020050306. PMID 9833102